CLINICAL TRIAL: NCT01158339
Title: Dare to Move: Treatment of Movement Phobia in Patient With Low Back Pain A Randomized Controlled Study of Two Methods Comparing the Role of Exposure in Session
Brief Title: Dare to Move: Treatment of Movement Phobia in Patient With Low Back Pain
Acronym: Ryggbra
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Helse Nord-Trøndelag HF (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REK No 2010/48-2
Record Dates: First submitted 2010-05-21; First posted 2010-07-08 (Estimated); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Low Back Pain
Keywords: Low back pain; Cognitive behavioural therapy; Group therapy; Exposure in session
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: CBGT (Active Comparator): Cognitive Behavioural Group Therapy (CBGT)
  Interventions: Behavioral: Arm 1: CBGT
- Arm 2: CBGT-ISE (Experimental): Cognitive Behavioural Group Therapy, with in-Session Exposure (CBGT-ISE).
  Interventions: Behavioral: Arm 2: CBGT-ISE

INTERVENTIONS:
Behavioral: Arm 2: CBGT-ISE — Intervention with active performance of the feared movements during group sessions.
  Arms: Arm 2: CBGT-ISE
Behavioral: Arm 1: CBGT — Intervention according to previously mentioned methods.
  Arms: Arm 1: CBGT

SUMMARY:
Unspecific low back pain (LBP) is a major world wide health problem. The purpose of this study is to improve the care of LBP.

Our hypothesis is that Cognitive Behavioural Therapy (CBT) with physical intervention during group sessions focusing on fear and avoidance behaviour will be more effective than physical therapy alone.

The study has two arms. Both will receive education related to LBP and appropriate advice regarding how to react and behave towards their LBP.

The main focus in the intervention group will be:

* Identifying their fear of movements and perform the frightened movements during the group sessions.
* Reassuring that gradually normalizing daily activities will not be harmful but rather reduce their pain.

DETAILED DESCRIPTION:
Cognitive-behavioural treatment is the treatment of choice in the treatment of most patients with chronic LBP. Several randomized controlled trials and recent meta-analysis have demonstrated the potent effects of CBT.

The fear and avoidance model developed by Vlaeyen and Linton has been recommended to be applied in the treatment of patients with chronic low back pain. No randomized controlled study has been published comparing the use of a fear and avoidance treatment with a comparison treatment. Such a study is highly warranted to examine if the model actually has a superior effect compared to other CBT-based treatments. In addition, it is of vital importance to examine whether all patients profit better from such a treatment or whether it only will demonstrate superior effect in a subgroup of patients with chronic low back pain.

PROBLEMS OF INTEREST:

Main aims are to improve the treatment of patients with chronic LBP by:

* 1) Testing the effect of a treatment assumed by the international scientific community to be the treatment of choice;
* 2) To develop a diagnostic screening procedure that at an initial examination can differentiate patients that need special treatment attention in the form of exposure towards feared movements from those who can benefit sufficiently from just receiving appropriate advice.
* 3) To identify the mechanism of change in the treatment of LBP.

METHODS:

Subjects will be recruited from general practitioners in the county of Nord-Trøndelag and from our department.

The study is clinical prospective and randomized. Each session will be videotaped. Two independent raters will rate three random sessions from both the intervention and non-intervention groups. Treatment differentiability will be measured by assessing the amount of time (minutes) spent exposing the patients to various movements in the session (ISE). According to the manuals, amount of ISE in CBGT (cognitive Behavioural Group Therapy) should be zero and between ten to twenty minutes in the CBGT-ISE (cognitive Behavioural Group Therapy- In Session Exposure) condition.

In addition, in both groups the therapists conducting the treatments are instructed to measure amount of time devoted to ISE in each session.

The therapist will rate every session. Three out of six sessions will also be timed and rated by two independent raters. The consistency of the time measured by the therapist and the independent raters will be compared in order to assure correctness of reported time spent in session. The raters will also asses the quality of the sessions. If the ratings are consistent across therapists and independent raters, a total ISE score for each treatment group will be computed.

THE TWO ARMS:

Arm 1: CBGT Patients will be given a manualised group treatment based on a fear and avoidance model. A main focus will be identifying fear of movements. The patients will in a spoken manner be reassured that they gradually can begin to perform normal daily activities and perform movements in a normal manner without using various forms of safety behaviours. Dysfunctional thinking patterns will be identified and challenged. Ten to twenty minutes of each session will be devoted to reassuring patients that various forms of feared movements can be performed in a graded fashion based on a feared hierarchy.

Arm 2: CBGT-ISE Patients will be given a manualised group treatment based on a fear and avoidance model. A main focus will be identifying fear of movements. The patients will in a spoken manner be reassured that they gradually can begin to perform normal daily activities and perform movements in a normal manner without using various forms of safety behaviours. Dysfunctional thinking patterns will be identified and challenged.

Ten to twenty minutes of each session will be devoted to actually exposing the patients to various feared movements and performing these in a graded fashion based on a fear hierarchy.

ELIGIBILITY:
Inclusion Criteria:

* Low Back Pain (LBP) lasting from 3 months to 10 years.
* Pain of such a severity that life of quality is reduced.
* The patient's main problem must be LBP, localized from L1 to S1.
* The pain must not be caused by nerve root affection (e.g. herniated disc)
* The patient has to be able to understand instructions given in Norwegian and to take part in a group activity.
* The patient must be partly or fully on sick leave from work.
* The patient must have a regular work to return to.

Exclusion Criteria:

* 100 % disability pension, of any reason.
* LBP that clearly is secondary to other somatic or psychiatric disorders.
* Alcohol and drug abuse.
* LBP caused by ankylosing spondylitis and other spondylarthropathies.
* Patients with "red flags" such as bladder- and anal paresis, impotence or progressing paresis.
* Ongoing insurance affairs for all types of sickness, injuries and accidents both against insurance companies and NAV (The Norwegian Labour and Welfare Administration)
* Indication for back surgery or performed back surgery last 12 months
* On medication known to cause depression or other psychiatric symptoms

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Absenteeism from work | Week 52
  Registrations of absenteeism will be given by the Norwegian Sick leave Register. This has certainly to be retrospectively (Is already approved)

SECONDARY OUTCOMES:
Pain | Will be done the following weeks: -1., 6., 14., and 52.
  Pain. Pain Brief Inventory
Physical functioning. | Will be done the following weeks: -1., 6., 14., and 52.
  Physical functioning: SF-8 health survey
  Will be done the following weeks: -1., 6., 14., and 52.
Emotional functioning | Will be done the following weeks: -1., 6., 14., and 52.
  Emotional functioning: Beck Depression Inventory
Patient ratings of improvement and satisfaction with treatment | Will be done the following weeks: -1., 6., 14., and 52.
  Questionaire
Health-related quality of life | Will be done the following weeks: -1., 6., 14., and 52.
  Questionaire
Coping/catastrophising | One week before intervention starts, then week 2 during the intervention, week 6 after finished intervention, week 14 after the booster and week 52.
  Other symptoms and adverse events during treatment Patient disposition and characteristics data
Side effects | Will be done the following weeks: -1., 6., 14., and 52.
  Any types. Drugs are not at all introduced in the study
Quality of life | Will be done the following weeks: -1., 6., 14., and 52.
  Health-related quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Tore Charles Stiles, prof, Study Director — Norwegian University of Science and Technology
Locations (1):
- Levanger Hospital, Levanger, Norway

REFERENCES:
- [Result] Ryum T, Hartmann H, Borchgrevink P, de Ridder K, Stiles TC. The effect of in-session exposure in Fear-Avoidance treatment of chronic low back pain: A randomized controlled trial. Eur J Pain. 2021 Jan;25(1):171-188. doi: 10.1002/ejp.1659. Epub 2020 Oct 6. PMID 32964624